CLINICAL TRIAL: NCT05645601
Title: Early Clinical Study of Allogenic CAR-NK Targeted CD19 (JD010) in the Treatment of Adult Relapsed or Refractory B-cell Malignancies
Brief Title: CAR-NK Targeted CD19 for r/r B-cell Malignancies
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Affiliated Hospital to Academy of Military Medical Sciences (Other)
Collaborators: Beijing JD Biotech Co. LTD. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAR-NK-JD010
Record Dates: First submitted 2022-12-01; First posted 2022-12-09 (Actual); Last update posted 2022-12-09 (Actual); Status verified 2022-12

CONDITIONS: Adult Relapsed/Refractory B-cell Hematologic Malignancies
MeSH Terms: conditions — Recurrence

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CD19 CAR-NK(JD010) (Experimental): CD19-CAR-NK is an allogenic CD19-Targeted chimeric antigen receptor NK-cell (CAR-NK) therapy.
  Interventions: Biological: CD19-CAR-NK

INTERVENTIONS:
Biological: CD19-CAR-NK — The relapsed/refractory B-cell hematologic malignancies patients will receive FC (F, Fludarabine, C, Cyclophosphamide) chemotherapy followed by 3 infusions of JD010 cells up to 2 dose levels (5x10^6/kg, 2x10^7/kg) after FC chemotherapy.

SUMMARY:
This is a single-centre, single-arm and open-label study to investigate the safety and efficacy of JD010 in adult patients with relapsed or refractory B cell hematologic malignancies. JD010 injection is a CD19-targeted chimeric antigen receptor modified natural killer cells (CAR-NK) derived from a healthy donor

ELIGIBILITY:
Inclusion criteria:

1. Age ≥ 18 years old, no gender or race;
2. Expected survival period ≥ 3 months;
3. Eastern Cooperative Oncology Group (ECOG) performance status score of 0 to 2;
4. Confirmed relapsed/refractory B-cell malignancies and tumor cells expressing CD19;
5. Adequate organ function:

   A. Liver function: ALT≤3×ULN, AST≤3×ULN, total bilirubin≤2×ULN; B. Coagulation function: international normalized ratio (INR) or activated partial thromboplastin time (APTT) ≤ 1.5×ULN; C. Renal function: serum creatinine≤1.5×ULN or creatinine clearance rate ≥30mL/min; D. Cardiac function: Left ventricular ejection fraction (LVEF) ≥ 50%;
6. Women of child-bearing potential and all male participants must use effective methods of contraception for at least 12 months after infusion.;
7. Informed Consent/Assent: All subjects must have the ability to understand and the willingness to sign a written informed consent.

Exclusion Criteria:

1. Central nervous system involved;
2. Known contraindication to the protocol defined lymphodepleting chemotherapy regimen of fludarabine/cyclophosphamide;
3. Systemic use of hormones within 4 weeks prior to enrollment (except for patients with inhaled corticosteroids);
4. Any active infection requiring systemic therapy by intravenous infusion within 14 days prior to the first dose of study drug, including: HBV, HCV, HIV, syphilis infection, or active pulmonary tuberculosis.
5. History of hypersensitivity reactions to murine protein-containing products, or macromolecular biopharmaceuticals such as antibodies or cytokines;
6. Patients cannot guarantee effective contraception (condom or contraceptives, etc.) within 1 years after enrollment;
7. Women who are pregnant (urine/blood pregnancy test positive) or lactating;
8. Suffering from a serious autoimmune disease or immunodeficiency disease; 9 Suffering from mental illness;

10. Known alcohol dependence or drug dependence; 11. According to the investigator's judgment, the patient has other unsuitable grouping conditions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2024-05-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicities (DLTs) | 1 Months
Treatment-related adverse events | 3 months
Objective Response Rate (ORR) | 3 months

SECONDARY OUTCOMES:
Progression free survival (PFS) | 12 months
Overall Survival (OS) | 12 months
Proportion of subjects with minimal-residual disease (MRD) negative response | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- The Fifth Medical Center of Chinese People's Liberation Army (PLA) General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No